CLINICAL TRIAL: NCT06001983
Title: Effects of Imaginary Resisted Exercises Versus Physical Resisted Exercises on Hand Grip Strength in Children With Hemiplegic Cerebral Palsy
Brief Title: Effect of Imaginary Resisted Therapy Versus Physical Resisted Therapy on Hemiplegic Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0721
Record Dates: First submitted 2023-06-14; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Hemiplegic Cerebral Palsy
Keywords: Hemiplegic Cerebral Palsy, Hand Grip Strength, Imaginary Resisted Exercises, Physical Resisted Exercises.

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Imaginary resisted exercises (Experimental): • Handgrip exercises with the imagination of resistance in hand by getting feedback in VR Box will be given as an intervention. Stretching will be given at the beginning and the end of each session. This will include imaginary resistance exercises for handgrip by using Virtual Reality Box. Five types of different resistances will be imagined by patients by watching their own videos in VR box, which will be recorded on day one to make them familiar with the resistive objects and the resistance experienced from them by asking patients to perform 15-15 repetitions of each object. Every imaginary resistance exercise will have 15 repetitions. After performing exercises, the participants will ask to perform Finger-to-Nose Test and Purdue Pegboard Test.
  Interventions: Other: imaginary resisted exercises
- Physical resisted exercises (Experimental): Handgrip exercises with physical resistance in hand will be given as an intervention. Stretching will be given at the beginning and the end of the session. 5 different types of resistances will be given to patients for making themselves familiarize themselves with the type of resistance applied by each object, that they will experience in further sessions, by asking them to perform 15-15 repetitions of each object. Every physical resistance exercise will have 15 repetitions. After performing exercises, the participants will ask to perform Finger-to-Nose Test and Purdue Pegboard Test. In physical resistance exercises, resistive force is applied to the targeted region by using different and appropriate resistive objects
  Interventions: Other: physical resisted exercises

INTERVENTIONS:
Other: imaginary resisted exercises — 1. Imagination of squeezing a Sponge ball 15 reps
  2. Imagination of Finger Exerciser 15 reps
  3. Imagination of Theraband 15 reps
  4. Imagination of pressing Rubber ball 15 reps
  5. Imagination of pressing Hard object 15 reps
  Arms: Imaginary resisted exercises
Other: physical resisted exercises — 1. Resisted exercise of Squeezing a Sponge ball 15 reps
  2. Resisted exercise of Finger Exerciser 15 reps
  3. Resisted exercise of pulling theraband 15 reps
  4. Resisted exercise of pressing Rubber ball 15 reps
  5. Resisted exercise of pressing Hard object 15 reps
  Arms: Physical resisted exercises

SUMMARY:
The purpose of this study is to compare the effects of imaginary resisted exercises versus physical resisted exercises on hand grip strength in hemiplegic cerebral palsy

DETAILED DESCRIPTION:
Cerebral palsy (CP) is one of the most frequent causes of motor disability in children. CP is a group of permanent disorders of the development of movement and posture, causing activity limitations that are attributed to non-progressive disturbances that occurred in the developing fetal or infant brain. The risk factors for CP can be divided into pre-conception, prenatal, perinatal and postnatal ones. Twenty five percent of children with CP have spastic hemiplegia. Hemiplegic cerebral palsy falls in anatomic classification of cerebral palsy which affects only one side of body. Children who have hemiplegic cerebral palsy have absolutely no use of one side of the body. This means their shoulder; arm, hand, leg and foot are all completely paralyzed. So, in order to improve strength in upper extremity and hand, resistance exercises are used.

The study will be a randomized control trial. Patients will be recruited into two groups using simple random assignment. Non probability convenient sampling will be used. Data will be collected from patients with hemiplegic cerebral palsy by using Jamar dynamometer which is consider as a gold standard in measuring repetitive gripping, goniometer for range of motion and Finger to nose test to access the upper extremity function in stroke patient Those who will meet the inclusion criteria will be recruited. Group A will receive imaginary resisted exercise therapy Five types of different resistances will be imagined by patients by watching their own videos in VR box, which will be recorded on day one to make them familiar with the resistive objects and the resistance experienced from them by asking patients to perform 15-15 repetitions of each object. Group B will receive physical resisted exercise therapy in which 5 different types of resistances will be given to patients for making themselves familiarize themselves with the type of resistance applied by each object, that they will experience in further sessions, by asking them to perform 15-15 repetitions of each object. Every physical resistance exercise will have 15 repetitions. At the end of each session patient will perform finger to nose test and Purdue peg board test. After collecting data from the defined setting, it will be entered and analyzed using statistical package for social sciences (SPSS) for Windows Software, version 21.

ELIGIBILITY:
Inclusion Criteria:

* Congenital infantile hemiplegia.
* Aged between 6 and 12 years.
* Lack of use of the affected upper limb.
* Level I-III of the Manual Ability Classification System (MACS).
* Students scoring of Modified Ashworth Scale should be 3 or less than 3 out of 5 for the same muscle groups of previously mentioned movements.

Exclusion Criteria:

* Low cognitive level compatible with attending a special education school.
* Presence of contractures in the affected upper limb affecting the functional movement.
* Surgery in the six months previously to the treatment.
* Botulinum toxin in the two months previously to or during the intervention.
* Pharmacologically uncontrolled epilepsy

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-09-20 (Estimated)

PRIMARY OUTCOMES:
Jamar Dynamometer (Hydraulic Hand Dynameter) | 4 weeks
  The Jamar is the primary outcome measure for assessing hand grip strength
Finger to Nose Test | 4 weeks
  It is a part of the Fugl-Meyer Assessment for upper extremity to evaluate impairment of upper limb in stroke patients. The total movement time is used as a clinical outcome measure for quantification of movement quality and motor performance. Most commonly the person is seated and upon command moves the index fingertip back and forth between the ipsilateral knee and the tip of the nose five times, as fast, as accurate, as possible
Purdue Peg Board Test | 4 weeks
  It is a functional assessment tool to screen for hand dexterity. It was designed to assess fine motor hand function using three common objects, pegs, washers, and collars, to be inserted on
  a pegboard. With its long history and wide usage, its reliability in healthy subjects is well established because it employs tasks that resemble activities of daily living. It is economical and easy to administer
Goniometer | 4 weeks
  Goniometer has been the most widely used tool for measuring joint range of motion. To ensure reliable measurement, standardized, specific positions and landmarks are used to measure each joint movement
Cell Phone Camera | 4 weeks
  Redmi Note 7 with front camera 13 MP or above and Rear camera 48 MP or above

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nosheen Manzoor, MS OMPT, Principal Investigator — Riphah International University
Locations (1):
- Govt. National special education centre, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No